CLINICAL TRIAL: NCT03504501
Title: Improvement of Synaptic Plasticity and Cognitive Function in RAS Pathway Disorders
Brief Title: Synaptic Plasticity and Cognitive Function in RASopathies
Acronym: SynCoRAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has been terminated prematurely due to recruitment difficulties. Current status: recruitment stopped and cleaning of the database is ongoing.
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SYN-1748-MAL-0030-I; 2016-005022-10 (EudraCT Number)
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-05

CONDITIONS: Impaired Synaptic Plasticity; Impaired Cognition
Keywords: RASopathies, neurofibromatosis type 1, noonan syndrome, synaptic plasticity, transcranial magnetic stimulation
MeSH Terms: conditions — Cognition Disorders; Neurofibromatosis 1; Noonan Syndrome | interventions — Lovastatin; Lamotrigine

STUDY DESIGN:
Intervention Model Description: Monocenter, randomized, double-blind, parallel-group, placebo controlled, cross-over design with a series of three experiments (Noonan Syndrome: 2 experiments; Neurofibromatosis type 1 1 experiment) and n=14 participants per experiments
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exp. I: Noonan Syndrome - Lovastatin (Experimental): 200 mg Lovastatin daily for four days / Lovastatin-placebo (cross-over) prior to transcranial magnetic stimulation and test of attentional performance
  Interventions: Drug: Lovastatin
- Exp. II: Noonan Syndrome - Lamotrigine (Experimental): 300 mg Lamotrigine single dose / Lamotrigine-placebo prior to transcranial magnetic stimulation and test of attentional performance
  Interventions: Drug: Lamotrigine
- Exp. III: Neurofibromatosis Type 1 - Lamotrigine (Experimental): 300 mg Lamotrigine single dose / Lamotrigine-placebo prior to transcranial magnetic stimulation and test of attentional performance
  Interventions: Drug: Lamotrigine

INTERVENTIONS:
Drug: Lovastatin — oral application prior to transcranial magnetic stimulation intervention
  Arms: Exp. I: Noonan Syndrome - Lovastatin
Drug: Lamotrigine — oral application prior to transcranial magnetic stimulation intervention
  Arms: Exp. II: Noonan Syndrome - Lamotrigine; Exp. III: Neurofibromatosis Type 1 - Lamotrigine

SUMMARY:
The project is targeting cognitive impairment, one of the main health problems of patients with RAS pathway disorders. The aim of this study is to translate findings of animal studies to humans. This has been done by the applicants successfully for Lovastatin in Nf1. This result will be transferred to patients with Noonan Syndrome. lamotrigine is most likely a more effective and promising substance improving synaptic plasticity and consecutive cognitive function. It is expected that both substances are improving synaptic plasticity as well as alertness and changes in alertness may be a precondition for improvement of cognition.

ELIGIBILITY:
Inclusion Criteria:

1. Group 1: NS, Group 2: NF1 (both genetically assured)
2. Age ≥16 years
3. The adolescent (≥16) and legal guardian who are capable to give their consent and understand the aim and rationale of the study. In case of doubts, an independent medical practitioner will evaluate the capacity to consent.
4. Signed informed consent if ≥ 16 years and legal guardian.
5. Persons who are ≥ 18 years old and capable to give their consent and understand the aim and rationale of the study. In case of doubts, an independent medical practitioner will evaluate the capacity to consent.
6. Signed informed consent if ≥ 18 years.
7. Male participants and female participants who are not capable of bearing children or who use a method of contraception that is medically approved by the health authority of the respective country.

Exclusion Criteria:

1. Epilepsy
2. Medication with known CNS effects
3. Severe mental retardation
4. Side effects during previous medication with and contraindications for LTG and/or LOV and/or TMS
5. Psychiatric diseases
6. Previous history of allergic reactions with LTG and LOV medications
7. Potentially unreliable patients
8. Patients who are not suitable for the study in the opinion of the investigator
9. Pregnancy (incl. positive urine pregnancy test)
10. Persons who are incapable of giving consent or do not understand the aim or rationale of the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2023-02-09 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Long-term potentiation (LTP)-like plasticity measured with transcranial magnetic stimulation (TMS) | 12 months
  Changes in peak-to-peak amplitudes of motor evoked potentials (MEP)

SECONDARY OUTCOMES:
Difference between the neuropsychological testing of attention (Test of attentional performance) after placebo and after medication (LTG and LOV) | 12 months
  Response time (seconds) for alertness, visual scanning, Go/no Go, Incompatibility
Differences in short interval cortical inhibition (SICI) after placebo and after medication (LTG and LOV) | 12 months
  Changes in SICI

OTHER OUTCOMES:
Assessment of safety: EMG recording during TMS evaluation | 12 months
  Safety

CONTACTS AND LOCATIONS:
Locations (1):
- Technical University Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mainberger F, Jung NH, Zenker M, Wahllander U, Freudenberg L, Langer S, Berweck S, Winkler T, Straube A, Heinen F, Granstrom S, Mautner VF, Lidzba K, Mall V. Lovastatin improves impaired synaptic plasticity and phasic alertness in patients with neurofibromatosis type 1. BMC Neurol. 2013 Oct 2;13:131. doi: 10.1186/1471-2377-13-131. PMID 24088225
- [Derived] Jung NH, Egert-Schwender S, Schossow B, Kehl V, Wahllander U, Brich L, Janke V, Blankenstein C, Zenker M, Mall V. Improvement of synaptic plasticity and cognitive function in RASopathies-a monocentre, randomized, double-blind, parallel-group, placebo-controlled, cross-over clinical trial (SynCoRAS). Trials. 2023 Jun 6;24(1):383. doi: 10.1186/s13063-023-07392-z. PMID 37280688